CLINICAL TRIAL: NCT05815173
Title: Phase I/II Study of Ladarixin and Sotorasib in Advanced KRAS G12C Mutant Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Ladarixin With Sotorasib in Advanced NSCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-00959
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced Non-small Cell Lung Cancer With KRAS G12C Mutation
MeSH Terms: interventions — sotorasib; 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced NSCLC Patients (Experimental): Patients with KRASG12C mutant NSCLC will receive ladarixin and sotorasib in combination.
  Interventions: Drug: Sotorasib; Drug: Ladarixin

INTERVENTIONS:
Drug: Sotorasib — Sotorasib administered at the approved dose of 960mg PO once daily over 21-day treatment cycles.
Drug: Ladarixin — Ladarixin dose will be escalated as follows in Phase I: 3 patients will receive a starting dose of 200mg. If 2 or more patients experience a DLT at the lowest dose, the study will stop. If 0 out of 3 patients experience a DLT within 28 days, the next 3 patients will receive 300mg. If 1 out of 3 patients experiences a DLT, 3 more patients will be added to the 200 mg dose. If no more patients experience a DLT at 200mg, the next 3 patients will receive 300mg. If 2 of 6 patients receiving 200mg experience a DLT, the study will stop. If 2 or more patients experience DLTs, the maximum tolerated dose (MTD) will be the previous dose level. The same process will be repeated at each dose level. There will be 6 patients enrolled at MTD level for a maximum of 12 patients in the phase I cohort. Ladarixin will be administered as a twice-daily dose over a 21 day treatment cycle.
  In Phase II, ladarixin will be administered twice-daily at the recommended phase II dose over 21-day cycles.

SUMMARY:
This is a phase I/II, open-label, study of twice-daily oral ladarixin with sotorasib in participants with advanced KRASG12C mutant non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This study will enroll patients with KRASG12C mutant NSCLC not previously treated with KRASG12C inhibitors. Patients in this study will receive ladarixin and sotorasib. The primary objective of the Phase I portion is to define a recommended phase II dose (RP2D) of ladarixin when combined with sotorasib. The primary objective of the Phase II portion is to evaluate progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, according to local guidelines, signed and dated by the participant prior to the performance of any study-specific procedures, sampling, or analyses.
* Participant must be ≥18 years of age at the time of signature of the informed consent form (ICF).
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Histologically confirmed diagnosis of NSCLC (squamous or nonsquamous).
* Patients with metastatic or locally advanced NSCLC who are not candidates for curative surgery or curative radiation.
* Do not have an epidermal growth factor receptor (EGFR) mutation, anaplastic lymphoma kinase (ALK) translocation, rearranged during transfection (RET), ROS1 or other actionable molecular alterations that can be treated with FDA approved targeted agents.
* Patients must have documentation of presence of KRASG12C mutation in tumor tissue.
* Patients must have demonstrated progression of disease following treatment with anti-PD (L)-1 with or without platinum-based chemotherapy.
* Participants must have at least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Tumor lesions that have been irradiated ≥4 weeks before the start of treatment, and have subsequently had documented progression, may be chosen as target lesions in the absence of measurable lesions that have not been irradiated.
* Participants whose laboratory data at Screening meet the following criteria:

  * Absolute neutrophil count ≥1.5 × 109/L
  * Platelets ≥100 × 109/L
  * Hemoglobin ≥8 g/dL without transfusion within 7 days
  * Albumin ≥3 g/dL
  * Lymphocyte count ≥0.5 × 109/L
  * Serum bilirubin ≤1.5 × upper limit of normal (ULN), or ≤ 3.0 × ULN for subjects with Gilbert's Syndrome
  * AST and ALT ≤ 2x upper limit of normal (ULN)
  * International normalization ratio (INR) <1.5 if the patient is not on anticoagulants, or INR <3 after dose titration has been completed if the patient is on anticoagulants.
  * Renal clearance as estimated glomerular filtration rate (eGFR) by Modification of Diet in Renal Disease (MDRD) Study equation ≥50 mL/min/1.73m2.
* Persons of childbearing potential (POCBP, defined as a sexually mature person assigned female at birth) must have a negative serum pregnancy test prior to study entry. Women of non-childbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhea, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms), or have had surgical bilateral oophorectomy, hysterectomy, or bilateral tubal ligation >6 weeks prior to Screening.
* Persons assigned male at birth or persons assigned female at birth participants: Persons assigned male at birth participants with partners of childbearing potential and participants of childbearing potential are required to use 2 forms of acceptable contraception, including 1 barrier method, during their participation in the study and for 3 months following last dose. Persons assigned male at birth participants must also refrain from donating sperm during their participation in the study and for 12 months after the last dose of study medication.
* Participants must be able to swallow and retain orally administered medication.

Exclusion Criteria:

* History (≤1 years) or presence of hematological malignancies except stable CLL.
* History (≤1 years) of other cancer that is histologically distinct from the cancers under study, except for cervical carcinoma in situ, ductal carcinoma in situ, prostatic intraepithelial neoplasia, superficial non-invasive bladder tumors, or curatively treated stage I non-melanoma skin cancer.
* Known serious allergy to ladarixin, sotorasib, or excipients (e.g., microcrystalline cellulose).
* History (≤6 months before the start of treatment with the study drugs) of severe autoimmune disease (including ≥ Grade 3 or recurrent Grade 2 immune-related AEs of prior immuno-oncology therapy) or autoimmune disorder that requires chronic systemic corticosteroid treatment at immunosuppressive doses (prednisone >10 mg/day or equivalent).
* Brain or spinal metastases, except if treated by surgery or surgery plus radiotherapy or radiotherapy alone, with no clinical evidence of progression or hemorrhage for ≤7 days before the start of treatment with the study drugs, and has not received any systemic corticosteroids for ≥7 days before the start of treatment with the study drugs.
* History (≤6 months before the start of treatment with the study drugs) of pericarditis (any grade) or pericardial effusion (Grade ≥2).
* History of interstitial lung disease, radiation pneumonitis which required steroid treatment, idiopathic pulmonary fibrosis, drug-induced pneumonitis, idiopathic pneumonitis, or organizing pneumonia.
* Active infection requiring systemic treatment at the start of treatment in this trial. A washout period of 7 days after the last dose of antibiotics prior to first dose of study drug is required.
* History of seropositive status for human immunodeficiency virus (HIV) at any time before the start of treatment as determined by presence of anti-HIV-1 or anti-HIV-2 antibodies.

  -- Note: Testing for seropositive status during Screening will be at the discretion of the investigator in participants without previously reported results.
* Has active hepatitis B, or hepatitis C infection.

  * Note: Participants with hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA polymerase chain reaction (PCR) that is below the limit of detection) are permitted. Participants with controlled infections must undergo periodic monitoring of hepatitis B virus DNA.
  * Note: Participants who are hepatitis C virus antibody positive (HCV Ab+), who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) may be enrolled into the study. Participants with controlled infections must undergo periodic monitoring of HCV RNA per treating physician.
* History (≤6 months before the start of treatment) of any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the investigator and sponsor, could affect the patient's participation in the study such as:

  * Nonmalignant illnesses that are uncontrolled or whose control may be jeopardized by this study treatment.
  * Nonmalignant decompensated liver disease.
  * Significant gastrointestinal abnormalities or a chronic condition, including inability to swallow the formulated product, delayed gastric emptying, chronic active Crohn's disease that requires steroid therapy at any dose, refractory nausea and vomiting, and/or prior surgical procedures affecting absorption or requirement for intravenous alimentation.
* History (≤6 months before the start of treatment with the study drugs) of any of the following: acute myocardial infarction, unstable angina pectoris, coronary artery bypass graft, or cerebrovascular accident.
* Participants who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * Significant ventricular or supraventricular arrhythmias (patients with sinus arrhythmia or chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
  * Left ventricular ejection fraction (LVEF) <50% assessed by echocardiogram (ECHO) or multigated acquisition scan (MUGA) within 6 months before the start of treatment with the study drugs and at screening.
  * Resting bradycardia (<50 beats per minute) determined as the mean of 3 heart rate values from the screening triplicate 12-lead electrocardiograms (ECGs) obtained.
  * Other clinically significant heart disease such as congestive heart failure New York Heart Association Class II-IV.
* Participants with QT interval >470 msec at screening using Fridericia's formula (QTcF), determined as the mean of 3 QTcF values from the screening triplicate ECG.
* Known history (≤6 months before the start of treatment with the study drugs) of significant inflammatory eye disease, central serous retinopathy, uveitis, or evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndrome).
* Participants experiencing unresolved Grade >1 toxicity before the start of treatment with the study drug except for hair loss (alopecia), Grade 2 neuropathy is permitted if the investigator permits and written approval is granted by the medical monitor.
* Participants who have neuromuscular disorders that are associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis spinal muscular atrophy).
* History (≤6 months before the start of treatment with the study drugs) of malignant biliary obstruction, except for patients with a functioning biliary stent.
* Persons who are pregnant or breast-feeding.
* Has received or will receive a live vaccine within 30 days prior to the first administration of study medication. Seasonal flu vaccines that do not contain live vaccine are permitted.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Known or suspected hypersensitivity to the active pharmaceutical ingredient, non-steroidal anti-inflammatory drugs or any excipient of the investigational medicinal products (e.g. lactose and croscarmellose) as well as patients with congenital lactase deficiency, galactosaemia or glucose-galactose intolerance.
* History of treatment with KRAS inhibitors.
* History of an allogeneic bone marrow or solid organ transplant.
* Use of systemic anticancer agent (except for antiandrogen therapy for prostate cancer, therapy for bone metastases or cancer-related hypercalcemia) or investigational drug is prohibited ≤28 days for biologics and intravenous chemotherapy, or ≤14 days or 2 half-lives for small molecules, whichever is longer, prior to the first dose of ladarixin.
* History of radiation therapy ≤7 days prior to the first dose of ladarixin.
* Use of drugs known to be moderate or strong CYP3A4 inhibitors or inducers or sensitive CYP3A4 substrates with a narrow therapeutic index is prohibited ≤14 days before the start of treatment with the study drug until the end-of-treatment visit. Some of these medications may be allowed at the investigator's discretion after written approval by the medical monitor.
* Treatment with drugs metabolized by CYP2C9 with a narrow therapeutic index [i.e., phenytoin, warfarin, and high dose of amitriptyline (>50 mg/day)].
* Use of herbal drugs and supplements known to be moderate or strong CYP3A4 inhibitors or inducers or sensitive CYP3A4 substrates with a narrow therapeutic index is prohibited ≤14 days before the start of treatment with the study drug until the end- of-treatment visit. These herbal medications include but are not limited to: St. John's wort, cannabis (including "medical marijuana"), kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.
* History (≤28 days before the start of treatment with the study drugs) of major surgery or trauma or likelihood to require surgery at any time until the permanent discontinuation of treatment (the significance will be determined by the investigator after consultation with the medical monitor).
* Participants who start erythropoietin or G-CSF, pegfilgrastim, or filgrastim ≤2 weeks before start of treatment with the study drug.
* History (≤1 weeks before the first dose of ladarixin) of transfusion of whole blood, red blood cells or platelet packets.
* History (≤2 weeks before the start of treatment with the study drugs) of medications with known risk of Torsades de Pointes (cardiac arrhythmia due to drug-induced QTc prolongation).
* Use of H2-receptor antagonists, proton pump inhibitors, and/or intraluminal antacids within 3 days or 5 half-lives (whichever is longer) prior to starting ladarixin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) during 1st Treatment Cycle among Phase I Participants | Up to Day 21 (End Treatment Cycle 1, each cycle is 21 days)
  DLTs are defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Progression Free Survival (PFS) | Up to End of Survival Follow-Up (Up to Month 36)
  PFS is the amount of time (months) from initial treatment to disease progression or death from any cause.

SECONDARY OUTCOMES:
Percent of Participants who Experience Grade 5 Treatment-Related Adverse Events per CTCAE 5.0 | Up to End of Survival Follow-Up (Up to Month 36)
  Number of participants whose most severe treatment-related adverse event was rated Grade 5 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, where Grade 5 = death related to adverse event.
Percent of Participants who Experience Grade 4 Treatment-Related Adverse Events per CTCAE 5.0 | Up to End of Survival Follow-Up (Up to Month 36)
  Number of participants whose most severe adverse event related to treatment was rated Grade 4 according to CTCAE version 5.0, where Grade 4 = life-threatening consequences; urgent intervention indicated.
Percent of Participants who Experience Grade 3 Treatment-Related Adverse Events per CTCAE 5.0 | Up to End of Survival Follow-Up (Up to Month 36)
  Number of participants whose most severe treatment-related adverse event was rated Grade 3 according to CTCAE version 5.0, where Grade 3 = Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; or limiting self-care activities of daily living (ADL).
Percent of Participants who Experience Grade 2 Treatment-Related Adverse Events per CTCAE 5.0 | Up to End of Survival Follow-Up (Up to Month 36)
  Number of participants whose most severe treatment-related adverse event was rated Grade 2 according to CTCAE version 5.0, where Grade 2 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
Percent of Participants who Experience Grade 1 Treatment-Related Adverse Events per CTCAE 5.0 | Up to End of Survival Follow-Up (Up to Month 36)
  Number of participants whose most severe treatment-related adverse event was rated Grade 1 according to CTCAE version 5.0, where Grade 1 = Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
Percent of Participants who Experience Complete Response (CR) | Up to End of Survival Follow-Up (Up to Month 36)
  Percent of participants whose best response is a CR according to RECIST 1.1, where CR = disappearance of all target lesions.
Percent of Participants who Experience Partial Response (PR) | Up to End of Survival Follow-Up (Up to Month 36)
  Percent of participants who best response is a PR according to RECIST 1.1, where PR = at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Percent of Participants who Experience Unconfirmed Complete Response (UCR) | Up to End of Survival Follow-Up (Up to Month 36)
  Percent of participants who best response is a CR according to RECIST 1.1, but the response has not been confirmed.
Percent of Participants who Experience Unconfirmed Partial Response (PR) | Up to End of Survival Follow-Up (Up to Month 36)
  Percent of participants who best response is a PR according to RECIST 1.1, but the response has not been confirmed.
Overall Survival (OS) | Up to End of Survival Follow-Up (Up to Month 36
  OS is the amount of time (months) from initial treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Salman Punekar, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - NYU Langone Health, Garden City, New York
  - NYU Langone Health, Mineola, New York
  - NYU Langone Health, New Hyde Park, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: salman.punekar@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to salman.punekar@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.